CLINICAL TRIAL: NCT06779773
Title: A Non-interventional, Observational Study to Evaluate Treatment Patterns and Safety of Avacincaptad Pegol (ACP/IZERVAY™) in Routine Clinical Practice in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Study to Learn How Avacincaptad Pegol (Izervay™) is Used in Clinical Practice in People Who Have Geographic Atrophy
Status: Recruiting | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 3021-MA-3543
Record Dates: First submitted 2024-12-16; First posted 2025-01-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy; Macular Degeneration
Keywords: Avacincaptad Pegol; IZERVAY™; Treatment patterns; Safety; Functional Outcomes
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Izervay: Patients with geographic atrophy (GA) secondary to AMD who have made decision to begin treatment with Izervay
  Interventions: Drug: Avacincaptad pegol (ACP)

INTERVENTIONS:
Drug: Avacincaptad pegol (ACP) — intravitreal injection
  Other Names: IZERVAY™

SUMMARY:
This study is for people who have geographic atrophy due to age-related macular degeneration (AMD). AMD happens when the macula, the light-sensitive layer at the back of the eye called the retina, becomes damaged and causes a person's central vision to worsen. Geographic atrophy is an advanced form of AMD where cells in the retina waste away and die. Over time this can lead to permanent loss of vision.

Avacincaptad pegol can help slow down the worsening or progression of geographic atrophy. Avacincaptad pegol is a treatment approved in the US to treat geographic atrophy.

This study is about collecting information on how people with geographic atrophy are treated in routine clinical practice. This includes recording any medical problems from avacincaptad pegol. This is known as an observational study. Information will be collected from the peoples' medical records during and after treatment. The people in this study will have geographic atrophy in 1 or both eyes and they and their doctor has decided they will be treated with avacincaptad pegol. The individual's doctor decides on treatment, not the study sponsor (Astellas).

People that want to take part in the study will have eye examinations that they would usually have as part of their routine care. People will also be asked to complete surveys about their eye health. These surveys will occur when treatment starts and then every 6 months for the first 2 years. After 2 years the surveys will happen once a year. The people on the study can take part if their doctor provides treatment with avacincaptad pegol and they want to continue with the study. The people on the study can take part for up to 3 years or up to 5 years, depending on when they start the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) in 1 or both eyes
* Patient with a decision to treat with intravitreal avacincaptad pegol (ACP) prior to enrollment
* Patient willingness to complete the patient reported outcome (PRO).

Exclusion Criteria:

* Patients who have any contraindication or are not eligible for treatment with ACP, including the following:

  * Active ocular or peri-ocular infection in either eye
  * Active, suspected intraocular inflammation in either eye at enrollment/baseline visit
  * Hypersensitive to ACP or to any ingredient in the formulation
* Patients currently participating in an investigational program with interventions outside of routine clinical practice.
* Patients who have received ACP in the study eye. Note: Patients who have received or are receiving ACP in the fellow eye are eligible to be included in the study.
* Patients who have received any intravitreal complement inhibitor other than ACP in either eye. Note: Patients who have received an intravitreal complement inhibitor other than ACP in either eye and have completed the 90-day washout period are eligible to be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants from both academic and non-academic sites, urban and rural across the US to ensure a heterogenous population that is representative of the US GA secondary to AMD population and reflective of real-world practice patterns.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of ACP injections | Up to 61 Months
  The number of ACP injections.
Dose of ACP injection | Up to 61 Months
  The dose of each ACP injection.
Duration of treatment | Up to 61 Months
  The duration of treatment will be calculated as the difference between the date of the last injection and the date of the first injection plus 31 days (as the next injection would be expected at least 30 days after the last one).
Annual frequency of ACP injection | Up to 61 Months
  The annual frequency of ACP injections will be calculated as the total number of injections divided by the treatment duration in years.
Reasons for discontinuation of treatment with ACP | Up to 61 Months
  The reasons for discontinuation of treatment with ACP will be recorded.
Duration of the treatment interval | Up to 61 Months
  The treatment interval is defined as mean number of days between injections, if a study eye receives more than 1 injection.
Site characteristics | Day 1
  Characteristics of interest will be recorded including the type of setting (e.g., public/private facility, rural/urban).
Characteristics of patients with geographic atrophy (GA) secondary to AMD beginning treatment with Izervay | Day 1
  Characteristics of interest will be recorded.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 61 Months
  An AE is defined as any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal (investigational) product.
Number of participants with Serious Adverse Events (SAEs) | Up to 61 Months
  An SAE is defined as an AE that results in death, is life-threatening, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or other medically important events.
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to 61 Months
  TEAE is defined an AE observed after starting administration of the study drug and will continue until 30 days after the last administration or until last study visit, whichever is sooner.
Number of participants with Adverse Event of Special Interest (AESI) | Up to 61 Months
  AESIs are defined as the following AEs:
  * Endophthalmitis
  * choroidal neovascularization (CNV)
  * Intraocular inflammation (including retinal vasculitis)
  * Increased intraocular pressure (IOP) ≥ 30 mmHg at 30 minutes post injection deemed clinically significant by the investigator
  * Elevation of IOP post injection requiring surgical/procedural intervention
  * Ischemic optic neuropathy
Number of Participants maintaining vision | Up to 61 Months
  Maintaining vision is defined as not losing ≥ 15 letters on Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Time to vision loss using various thresholds | Up to 61 Months
  Time to vision loss is defined as the difference between the date when vision loss was reported for the first time and the start date of treatment.
Time to thresholds associated with ability to drive | Up to 61 Months
  Time to thresholds associated with the ability to drive will be based on visual acuity data captured as per standard of care.
Participant's reading speed | Up to 61 Months
  Reading speed will be captured as per standard of care and in the method determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (59):
- United States (59):
  - Phoenix Retina Clinical Trials, LLC, Phoenix, Arizona
  - Retinal Consultants of AZ, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - The Retina Partners, Encino, California
  - Harvard Eye Associates, Laguna Hills, California
  - Retina Consultants of Southern CA, Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Retina Macula Institute, Torrance, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Colorado Retina Associates, PLLC, Lakewood, Colorado
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Advanced Retina Institute, Bonita Springs, Florida
  - University of Miami, Coral Gables, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Eye Physicians of Pinellas PA dba Eye Institute of West Florida, Tampa, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - University Retina and Macula Associates, P.C., Oak Forest, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Cumberland Valley Retina Consultants,P.C., Hagerstown, Maryland
  - Retina Specialists, Towson, Maryland
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Retina Consultants of Minnesota PLLC, Saint Louis Park, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - Deep Blue Retina Clinical Research, Southaven, Mississippi
  - Eye Associates of North Jersey PA, Dover, New Jersey
  - NJ Retina, Edison, New Jersey
  - NJ Retina, Lakewood, New Jersey
  - Monmouth Retina Consultants, Little Silver, New Jersey
  - NJ Retina, Toms River, New Jersey
  - SightMD, Brentwood, New York
  - Retina-Vitreous Surgeons of Central NY, Liverpool, New York
  - NY Retina Ophthalmology PLLC, Massapequa, New York
  - Retina Associates of New York, New York, New York
  - Long Island Vitreoretinal Consultants, Scarsdale, New York
  - Vitreoretinal Consultants, Shirley, New York
  - North Carolina Retina Associates, Cary, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - The Ohio State University, Columbus, Ohio
  - CEI Physicians PSC, LLC dba, Dayton, Ohio
  - Verum Research, LLC, Eugene, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Mid South Retina Associates, Memphis, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina of North Texas, Dallas, Texas
  - Retina & Vitreous of Texas, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of Utah, P.C., Murray, Utah
  - Salt Lake Retina, Salt Lake City, Utah
  - The Retina Group of Washington, Fairfax, Virginia
  - Piedmont Eye Center, Inc., Lynchburg, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Retina & Vitreous Consultants of Wisconsin, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.